CLINICAL TRIAL: NCT00876746
Title: Optimization of Catheter Insertion Site for Continuous Peripheral Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Brian Ilfeld, M.D., M.S./ Principal Investigator, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Supra / Infra Catheters
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2009-04

CONDITIONS: Upper-extremity Surgery; Post-operative Pain
Keywords: Pain; surgery; catheter; nerve block; supraclavicular; infraclavicular; UCSD; moderate-to-severe pain; Supraclavicular catheter; Infraclavicular catheter
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Supraclavicular (Active Comparator): Patients will be randomized to placement of a nerve block in the supraclavicular position. After the catheter has been placed, sensory and motor deficit will be assessed and following surgery, for the next three days, the patient will be contacted by research staff to assess pain scores and other outcome measures.
  Interventions: Procedure: Supraclavicular vs. Infraclavicular ropivicaine infusion
- 2. Infraclavicular (Active Comparator): Patients will be randomized to placement of a nerve block in the infraclavicular position. After the catheter has been placed, sensory and motor deficit will be assessed and following surgery, for the next three days, the patient will be contacted by research staff to assess pain scores and other outcome measures.
  Interventions: Procedure: Supraclavicular vs. Infraclavicular ropivicaine infusion

INTERVENTIONS:
Procedure: Supraclavicular vs. Infraclavicular ropivicaine infusion — Patients will be randomized to one of two groups: nerve blocks in the supraclavicular location or the infraclavicular location. Following surgery the patient will be called by study staff to assess pain scores, sleep disturbances, infusion side effects, feeling in fingers and other study outcomes.

SUMMARY:
This research study is to determine if the insertion site of a perineural catheter or tiny tube placed next to the nerves that go to the part of the body (hand or arm) having surgery, affects the amount of pain relief that is experienced after surgery. Catheters will be placed in either the supraclavicular or infraclavicular location.

DETAILED DESCRIPTION:
To determine if a particular perineural local anesthetic catheter location (supraclavicular or infraclavicular) will maximize postoperative analgesia, minimize oral opioid requirements, minimize sleep disturbances resulting from postoperative pain, and maximize patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* unilateral, upper (at or distal to the elbow) extremity orthopedic surgery with moderate-to-severe postoperative pain expected
* patients already agree to and want a continuous brachial plexus block for postoperative analgesia

Exclusion Criteria:

* patients who have difficulty understanding the study protocol or caring for the infusion pump/catheter system
* patients who have any known contraindication to study medications
* insulin-dependent diabetes mellitus
* neuropathy of any etiology in the affected extremity
* contraindication to regional blockade (e.g. clotting deficiency)
* any known acute or chronic hepatic or renal insufficiency or failure
* any incision site outside of the catheter-effected area
* chronic opioid use
* history of opioid abuse
* obesity
* pregnancy
* incarceration
* inability to communicate with the investigators and hospital staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Surgical pain as measured on a 0-10 scale where 0=no pain and 10=worst imaginable pain. The values for the two different catheter locations will be compared to see which site is optimal for catheter placement. | 3 days

SECONDARY OUTCOMES:
Opioids consumed by patient each day after surgery as reported to study staff. | 3 days
Sleeping disturbances (difficulty sleeping and awakenings due to pain) as reported to the study staff. | 3 days
Infusion side effects (shortness of breath) as reported to study staff. | 3 day
Satisfaction with pain control as measured on a 0-10 scale where 0=very unsatisfied and 10=very satisfied, as reported to study staff at time of daily phone calls | 3 days
Sensory and motor deficits (ability to move fingers and numbness of fingers) as reported to study staff. | 3 days
Catheter site discomfort, leakage at catheter site, and catheter related pain on the 0-10 rating scale, where 0=no pain and 10=worst imaginable pain, as reported to study staff during phone calls. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States